CLINICAL TRIAL: NCT03806036
Title: The Effect Of Vitamin D Replacement Therapy On Serum Leptin And Follicular Growth Pattern In Women With Resistant Polycystic Ovarian Syndrome
Brief Title: The Effect Of Vitamin D Replacement Therapy On Serum Leptin And Follicular Growth Pattern In Women With Resistant Polycystic Ovary
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Maged, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 47
Record Dates: First submitted 2019-01-13; First posted 2019-01-16 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Vitamin D; Clomiphene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin D group (Active Comparator): 50 women will receive 300.000 I.U single dose of VIT D IM injection (Memphis company) , and in the next menstrual cycle induction done by clomiphen citrate 100mg daily for 5 days starting from third day of menstruation and HMG single dose on 8th day
  Interventions: Drug: Vitamin D; Drug: Clomiphene Citrate
- Control group (Placebo Comparator): 50 women will receive clomiphen citrate 100mg daily for 5 days starting from third day of menstruation and HMG single dose on 8th day
  Interventions: Drug: Clomiphene Citrate

INTERVENTIONS:
Drug: Vitamin D — 300.000 I.U single dose of VIT D IM injection
  Arms: Vitamin D group
Drug: Clomiphene Citrate — 100mg daily for 5 days starting from third day of menstruation
  Other Names: Clomid

SUMMARY:
The study included 100 female diagnosed with polycystic ovary syndrome. They were classified into 2 groups: Study group included 50 women will receive 300.000 I.U single dose of Vitamin D intramuscular injection (Memphis company) , and in the next menstrual cycle induction done by clomiphen citrate 100mg daily for 5 days starting from third day of menstruation and HMG single dose on 8th day . Control group included 50 women will receive only clomiphen citrate 100mg daily for 5 days starting from third day of menstruation and HMG single dose on 8th day. Serum 25 hydroxy Vitamin D3, Serum Leptin and FSH will be done to all women before and after intervention.

DETAILED DESCRIPTION:
The study included 100 female diagnosed with polycystic ovary syndrome diagnosed by by presence of 2 out of 3 criteria (according to ESHRE/ASRM in Rotterdam in 2003): oligoovulation and/or an ovulation , excess androgen activity (clinical or biochemical) and polycystic ovaries (by pelvic ultrasound "vaginal route").They were classified into 2 groups: Study group included 50 women will receive 300.000 I.U single dose of Vitamin D intramuscular injection (Memphis company) , and in the next menstrual cycle induction done by clomiphen citrate 100mg daily for 5 days starting from third day of menstruation and HMG single dose on 8th day . Control group included 50 women will receive only clomiphen citrate 100mg daily for 5 days starting from third day of menstruation and HMG single dose on 8th day. Serum 25 hydroxy Vitamin D3, Serum Leptin and FSH will be done to all women before and after intervention.

ELIGIBILITY:
Inclusion Criteria:

1- BMI: more than 25.0 kg/m2

2- PCO was diagnosed by presence of 2 out of 3 criteria (according to ESHRE/ASRM in Rotterdam in 2003)

1. oligoovulation and/or an ovulation
2. excess androgen activity (clinical or biochemical)
3. polycystic ovaries (by pelvic ultrasound "vaginal route")

3- Anovulatory patient resistant to induction with clomiphene citrate alone

Exclusion Criteria:

-1) BMI: more than 35.0 kg/m2

2) Infertile women due to any factor other than PCO

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2018-01-02 (Actual); Primary Completion 2019-02 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Ovulation | 14 days after menses
  appearance of dominant follicle 18 - 22 mm in diameter

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, Principal Investigator — Professor
Locations (1):
- Kasr Alainy medical school, Cairo, Egypt